CLINICAL TRIAL: NCT07147985
Title: Effects of Different Exercises on Energy Metabolism and Muscle Activation in Normal-Weight and Overweight Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanxi Normal University (Other)
Responsible Party: Principal Investigator, Haiwei Li, Professor, Shanxi Normal University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-0505
Record Dates: First submitted 2025-08-08; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-05

CONDITIONS: Energy Expenditure
Keywords: slow jogging; step frequency; energy expenditure; college students

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Step frequency group 1 (Experimental): Participants will receive step frequency in the following order:
  First test: 162 steps per minute; Second test: 180 steps per minute; Third test: 198 steps per minute.
  Interventions: Behavioral: 162 step frequency; Behavioral: 180 step frequency; Behavioral: 198 step frequency
- Step frequency group 2 (Experimental): Participants will receive step frequency in the following order:
  First test: 162 steps per minute; Second test: 198 steps per minute; Third test: 180 steps per minute.
  Interventions: Behavioral: 162 step frequency; Behavioral: 180 step frequency; Behavioral: 198 step frequency
- Step frequency group 3 (Experimental): Participants will receive step frequency in the following order: First test: 180 steps per minute; Second test: 162 steps per minute; Third test: 198 steps per minute.
  Interventions: Behavioral: 162 step frequency; Behavioral: 180 step frequency; Behavioral: 198 step frequency
- Step frequency group 4 (Experimental): Participants will receive step frequency in the following order:
  First test: 180 steps per minute; Second test: 198 steps per minute; Third test: 162 steps per minute.
  Interventions: Behavioral: 162 step frequency; Behavioral: 180 step frequency; Behavioral: 198 step frequency
- Step frequency group 5 (Experimental): Participants will receive step frequency in the following order:
  First test: 198 steps per minute; Second test: 162 steps per minute; Third test: 180 steps per minute.
  Interventions: Behavioral: 162 step frequency; Behavioral: 180 step frequency; Behavioral: 198 step frequency
- Step frequency group 6 (Experimental): Participants will receive step frequency in the following order:
  First test: 198 steps per minute; Second test: 180 steps per minute; Third test: 162 steps per minute.
  Interventions: Behavioral: 162 step frequency; Behavioral: 180 step frequency; Behavioral: 198 step frequency

INTERVENTIONS:
Behavioral: 162 step frequency — The exercise protocol lasted 21 minutes, comprising a 10-minute period of slow-pace running, preceded by a 3-minute quiet resting period and a 3-minute warm-up, and followed by a 5-minute recovery period after the warm-up and slow-pace running. 162 steps per minute crossover to 180 steps per minute and 198 steps per minute.
Behavioral: 180 step frequency — The exercise protocol lasted 21 minutes, comprising a 10-minute period of slow-pace running, preceded by a 3-minute quiet resting period and a 3-minute warm-up, and followed by a 5-minute recovery period after the warm-up and slow-pace running. 180 steps per minute crossover to 162 steps per minute and 198 steps per minute.
Behavioral: 198 step frequency — The exercise protocol lasted 21 minutes, comprising a 10-minute period of slow-pace running, preceded by a 3-minute quiet resting period and a 3-minute warm-up, and followed by a 5-minute recovery period after the warm-up and slow-pace running. 198 steps per minute crossover to 162 steps per minute and 180 steps per minute.

SUMMARY:
This clinical trial aims to investigate the effects of different exercise modalities on energy metabolism and muscle activation in both normal-weight and overweight university students.

The main question it aims to answer is:

Compared to normal-weight university students, does slow jogging at different step frequencies reduce body weight and increase energy expenditure (and metabolic rate) in overweight university students? Compared to normal-weight university students, does slow jogging at different step frequencies enhance muscle activation effects in overweight university students?

Researchers will compare three distinct step frequencies during slow jogging (162, 180, and 198 steps per minute) to determine which exercise modality is potentially more effective for increasing energy expenditure and metabolic rate.

Participants will:

Participants will sequentially undergo three separate testing sessions, each involving ultra-slow running at one of the three step frequencies (162, 180, or 198 steps per minute).

Testing sessions will occur once per week in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 23 years old;
2. BMI between 24.0 kg/m² and 27.9 kg/m² ;
3. No participation in any structured weight loss or weight control interventions (including exercise programs, pharmacological agents, or dietary regimens) within the preceding three months;
4. Cleared for exercise participation with no identified risks, as determined by the Physical Activity Readiness Questionnaire (PAR-Q);
5. Willing and able to comply fully with the experimental protocol, including completion of all training sessions and required measurements;
6. Provision of written informed consent.

Exclusion Criteria:

1. History of psychiatric disorders, diabetes mellitus, heart disease, hypertension, anemia, or any other contraindications to exercise (e.g., dizziness, chest pain, shortness of breath);
2. Immune dysfunction or severe hepatic or renal insufficiency;
3. Unhealthy habits, such as regular smoking or excessive alcohol consumption;
4. Current use of prescription medication (excluding contraceptives or incidental short-term medications, if specified and approved by the study investigators);
5. Coagulation disorders or a significant bleeding tendency.

Withdrawal and Termination Criteria:

1. Voluntary withdrawal from the study or discontinuation for any other reason;
2. Poor compliance, defined as failure to follow instructions or complete assigned tasks as required by the protocol;
3. Experiencing severe exercise intolerance or adverse reactions to the intervention.

Ages: 19 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Resting Energy Expenditure (REE) | Baseline
  Subjects abstained from strenuous activity, substances (medication/alcohol/caffeine), and smoking 24h pre-test; females avoided menstruation. Post 12h fast/sleep, subjects rested seated 15min. Resting HR measured (Polar RS400). Subjects fitted with cardiopulmonary telemetry (Cortex Metamax 3B), positioned supine. Maintained steady breathing, upward gaze, minimal movement. HR/V̇O₂ monitored until stabilization. 10min data collection; steady state = <5% V̇O₂ fluctuation over 5min.
Energy Expenditure at Step Frequencies | through study completion, an average of 4 weeks
  Telemetry/HR monitor worn for 3min warm-up. First test: 10min treadmill run (5 km/h) with HR/V̇O₂ recording. Two subsequent sessions followed. Randomized crossover prevented order effects: subjects drew lots for step frequency sequence (162, 180, 198 steps/min). Metronome ensured adherence.
Heart rate | through study completion, an average of 4 weeks
  Upon entering the laboratory, subjects wore a heart rate telemetry monitor (RS400 Polar, Finland) and rested seated for 15 minutes to obtain resting heart rate. Following warm-up, subjects commenced testing. A heart rate monitor was secured on the right wrist pre-exercise to continuously monitor heart rate during activity.
Electromyographic indicators | through study completion, an average of 4 weeks
  Wireless surface EMG data were acquired using the Trigno system (Delsys®, USA) at 2000 Hz. Electrodes were positioned at the mid-belly of each muscle parallel to the muscle fiber orientation. Signals were recorded from the:Biceps femoris、Rectus femoris、Tibialis anterior、Lateral gastrocnemius、Medial gastrocnemius. EMGworks Analysis® software (Delsys) processed raw signals.

SECONDARY OUTCOMES:
Post-Exercise Oxygen Consumption (EPOC) | through study completion, an average of 4 weeks
  EPOC was calculated from pre-/post-exercise oxygen consumption (O₂PRE/O₂POST) measured via portable cardiopulmonary telemetry (Cortex Metamax 3B): EPOC (L) = O₂POST (L) - O₂PRE (L) where: EPOC denotes excess post-exercise oxygen consumption, O₂POST represents post-exercise oxygen consumption, and O₂PRE represents pre-exercise oxygen consumption.
Fat Oxidation | through study completion, an average of 4 weeks
  Fat Oxidation Data were collected and analyzed using the portable cardiopulmonary telemetry system (Cortex Metamax 3B, Germany). The fat oxidation rate was calculated as follows: Fat oxidation rate (g/min) = ② Fat Oxidation Fat oxidation rate was derived as: 1.695 × V̇O₂ (L/min) - 1.701 × V̇CO₂ (L/min) (g/min) using mean V̇O₂/V̇CO₂ from final 2min of each stage. ③ Carbohydrate Oxidation Carbohydrate oxidation rate was calculated as: 4.585 × V̇CO₂ (L/min) - 3.226 × V̇O₂ (L/min) (g/min) using mean V̇O₂/V̇CO₂ from final 2min of each stage. All data collected/analyzed with Cortex Metamax 3B system.
Carbohydrate Oxidation | through study completion, an average of 4 weeks
  Carbohydrate oxidation rate was calculated as: 4.585 × V̇CO₂ (L/min) - 3.226 × V̇O₂ (L/min) (g/min) using mean V̇O₂/V̇CO₂ from final 2min of each stage. All data collected/analyzed with Cortex Metamax 3B system.
RPE | through study completion, an average of 4 weeks
  Immediately after each exercise stage, subjects rated perceived exertion using the Borg RPE scale. The 15-point scale (6-20; 6 = no exertion, 20 = maximal exertion) was administered and recorded post-stage.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi Normal University, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No